CLINICAL TRIAL: NCT05346289
Title: Elective Treatment Rates Among Patients With Intact Abdominal Aortic Aneurysms -Patient- and Aneurysm-related Factors as Determinants of Surgical Non-eligibility in Women and Men
Brief Title: Elective Treatment Rates and Surgical Non-eligibility Among Men and Women With Intact Abdominal Aortic Aneurysms
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Medical University of Graz (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Rebecka Hultgren, Prof., Senior Consultant, Karolinska University Hospital
Other Study IDs: ESPN201689310422
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Abdominal Aortic Aneurysm; Abdominal Aortic Aneurysm Without Rupture; Aneurysm; Aortic Aneurysm; Aneurysm Abdominal
Keywords: Sex differences; Elective treatment rate; Surgical eligibility; Surgical treatment; Conservative treatment; Untreated
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm; Aortic Aneurysm | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women
  Interventions: Procedure: Elective surgery for intact AAA
- Men
  Interventions: Procedure: Elective surgery for intact AAA

INTERVENTIONS:
Procedure: Elective surgery for intact AAA — Elective surgery including the following modalities: open repair, endovascular repair (EVAR), fenestrated end-vascular repair (FEVAR).

SUMMARY:
The overall aim is to determine the frequency by which women and men with intact abdominal aortic aneurysms (AAA) are treated with elective surgery at three vascular outpatient clinics in Europe, and to investigate whether the reasons to refrain from elective surgery differ between the sexes.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) is a local widening of the infrarenal aorta (1). The natural history of AAA is progressive and may lead to rupture, a true surgical emergency with a mortality rate of 100% without immediate treatment. Men are more commonly affected (2, 3), however, women demonstrate a notably elevated risk of rupture (4, 5) and constitute up to 1/3 of all ruptures (4, 5). One plausible explanation could be a sex discrepancy in elective treatment rates.

There is both national and international evidence implying that AAA treatments, both elective and emergent, are withheld among women (6-14). Studies on elective treatment rates are especially scarce, as the vast majority of databases and vascular registries only include data on treated AAA patients. A few single-center studies from the UK (6, 7, 15) and one meta-analysis (8) have recorded lower treatment rates among women. We have recently analyzed the issue of elective treatment rates in our group using a population-based approach (manuscript submitted). Of all patients diagnosed with an intact AAA in Sweden during 2001-2015 (n=32 393, 21% women), a crude proportion as high as 60 % did not proceed to receive surgical treatment. The proportion of untreated women (67 %) surpassed that of men (59 %). In the multivariate analyses, female sex and advanced age emerged as the strongest predictors for remaining untreated despite other characteristics such as comorbidities, civil status and individual disposable household income. The median time from diagnosis to treatment for those treated was surprisingly short at 1.6 years.

The foremost intention-to-treat variable that determines the indication for elective surgery is the maximal diameter of the aneurysm (55 mm in men, 50 mm in women; (16, 17)). Population-based investigations, while comprehensive, fall short in terms of aneurysm-specific data. Therefore, these analyses assume comparable diameter distributions and similar morphology for men and women. Similarly, longitudinal follow-up data from the clinical setting, such as records of patient's wishes and physiological preoperative examinations, cannot be extracted for the purpose of nationwide analyses. Thus, the question remains whether the observed gender gap in elective treatment rates persists after detailed considerations of patient- and aneurysm-specific characteristics. A discrepancy in elective treatment rates could also lead to different long-term outcomes, with higher rupture and mortality rates among women.

ELIGIBILITY:
Inclusion Criteria:

• Intact abdominal aortic aneurysm 30 mm or larger in men and women irrespective of underlying pathogenesis (atherosclerotic, mycotic, previous dissection).

Exclusion Criteria:

* Previous aortic surgery or surgical treatment for AAA
* Ruptured AAA at index contact

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All men and women diagnosed with an intact abdominal aortic aneurysm (ICD10 classification I71.4) and who fulfill the inclusion diameter criterion and none of the exclusion criteria are consecutively included from January 2014 and onwards at three vascular outpatient departments in Europe (Karolinska University Hospital, Stockholm, Sweden; St. Olav Hospital, Trondheim, Norway; Medical University of Graz, Graz, Austria) until reaching prespecified study target size according to power calculation (200 women, 200 men).
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Final Elective Treatment Status | End of follow-up in December 2021 with maximal possible follow-up of seven years.
  Relative frequency of women and men that were electively treated or left untreated, the latter group subcategorized into patients who did or did not reach the diameter threshold for surgical treatment (50 mm women, 55 men).
Sex-Specific Reasons for Remaining Untreated | Evaluated at the time of the conservative treatment decision during maximal follow-up of seven years.
  Frequency distribution of underlying reasons behind non-treatment among those men and women who reached the treatment threshold. Primary reason registered as patient- (comorbidity, patient's wish) or AAA-related (morphology).

SECONDARY OUTCOMES:
Rupture Rate | Study end December 2021.
  Sex-specific rates of rupture in each treatment arm during follow-up.
Mortality Rate | Study end December 2021.
  Sex-specific rates of mortality in each treatment arm during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sakalihasan N, Michel JB, Katsargyris A, Kuivaniemi H, Defraigne JO, Nchimi A, Powell JT, Yoshimura K, Hultgren R. Abdominal aortic aneurysms. Nat Rev Dis Primers. 2018 Oct 18;4(1):34. doi: 10.1038/s41572-018-0030-7. PMID 30337540
- [Background] Lederle FA, Johnson GR, Wilson SE; Aneurysm Detection and Management Veterans Affairs Cooperative Study. Abdominal aortic aneurysm in women. J Vasc Surg. 2001 Jul;34(1):122-6. doi: 10.1067/mva.2001.115275. PMID 11436084
- [Background] Scott RA, Bridgewater SG, Ashton HA. Randomized clinical trial of screening for abdominal aortic aneurysm in women. Br J Surg. 2002 Mar;89(3):283-5. doi: 10.1046/j.0007-1323.2001.02014.x. PMID 11872050
- [Background] Sweeting MJ, Thompson SG, Brown LC, Powell JT; RESCAN collaborators. Meta-analysis of individual patient data to examine factors affecting growth and rupture of small abdominal aortic aneurysms. Br J Surg. 2012 May;99(5):655-65. doi: 10.1002/bjs.8707. Epub 2012 Mar 5. PMID 22389113
- [Background] Brown LC, Powell JT. Risk factors for aneurysm rupture in patients kept under ultrasound surveillance. UK Small Aneurysm Trial Participants. Ann Surg. 1999 Sep;230(3):289-96; discussion 296-7. doi: 10.1097/00000658-199909000-00002. PMID 10493476
- [Background] Karthikesalingam A, Nicoli TK, Holt PJ, Hinchliffe RJ, Pasha N, Loftus IM, Thompson MM. The fate of patients referred to a specialist vascular unit with large infra-renal abdominal aortic aneurysms over a two-year period. Eur J Vasc Endovasc Surg. 2011 Sep;42(3):295-301. doi: 10.1016/j.ejvs.2011.04.022. Epub 2011 May 14. PMID 21576025
- [Background] Whittaker JD, Meecham L, Summerour V, Khalil S, Layton G, Yousif M, Jennings A, Wall M, Newman J. Outcome after Turndown for Elective Abdominal Aortic Aneurysm Surgery. Eur J Vasc Endovasc Surg. 2017 Nov;54(5):579-586. doi: 10.1016/j.ejvs.2017.07.023. Epub 2017 Sep 2. PMID 28874329
- [Background] Sweeting MJ, Masconi KL, Jones E, Ulug P, Glover MJ, Michaels JA, Bown MJ, Powell JT, Thompson SG. Analysis of clinical benefit, harms, and cost-effectiveness of screening women for abdominal aortic aneurysm. Lancet. 2018 Aug 11;392(10146):487-495. doi: 10.1016/S0140-6736(18)31222-4. Epub 2018 Jul 26. PMID 30057105
- [Background] Zommorodi S, Bottai M, Hultgren R. Sex differences in repair rates and outcomes of patients with ruptured abdominal aortic aneurysm. Br J Surg. 2019 Oct;106(11):1480-1487. doi: 10.1002/bjs.11258. Epub 2019 Aug 12. PMID 31403186
- [Background] Aber A, Tong TS, Chilcott J, Thokala P, Maheswaran R, Thomas SM, Nawaz S, Walters S, Michaels J. Sex differences in national rates of repair of emergency abdominal aortic aneurysm. Br J Surg. 2019 Jan;106(1):82-89. doi: 10.1002/bjs.11006. Epub 2018 Nov 5. PMID 30395361
- [Background] Kuhnl A, Erk A, Trenner M, Salvermoser M, Schmid V, Eckstein HH. Incidence, Treatment and Mortality in Patients with Abdominal Aortic Aneurysms. Dtsch Arztebl Int. 2017 Jun 5;114(22-23):391-398. doi: 10.3238/arztebl.2017.0391. PMID 28655374
- [Background] McPhee JT, Hill JS, Eslami MH. The impact of gender on presentation, therapy, and mortality of abdominal aortic aneurysm in the United States, 2001-2004. J Vasc Surg. 2007 May;45(5):891-9. doi: 10.1016/j.jvs.2007.01.043. Epub 2007 Mar 28. PMID 17391899
- [Background] Dueck AD, Johnston KW, Alter D, Laupacis A, Kucey DS. Predictors of repair and effect of gender on treatment of ruptured abdominal aortic aneurysm. J Vasc Surg. 2004 Apr;39(4):784-7. doi: 10.1016/j.jvs.2003.10.064. PMID 15071441
- [Background] Katz DJ, Stanley JC, Zelenock GB. Gender differences in abdominal aortic aneurysm prevalence, treatment, and outcome. J Vasc Surg. 1997 Mar;25(3):561-8. doi: 10.1016/s0741-5214(97)70268-4. PMID 9081139
- [Background] Scott SW, Batchelder AJ, Kirkbride D, Naylor AR, Thompson JP. Late Survival in Nonoperated Patients with Infrarenal Abdominal Aortic Aneurysm. Eur J Vasc Endovasc Surg. 2016 Oct;52(4):444-449. doi: 10.1016/j.ejvs.2016.05.008. Epub 2016 Jun 30. PMID 27374814
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Background] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Derived] Talvitie M, Aldstedt-Nyronning L, Stenman M, Roy J, Cohnert T, Hultgren R. Women with large intact abdominal aortic aneurysms remain untreated. J Vasc Surg. 2023 Sep;78(3):657-667.e5. doi: 10.1016/j.jvs.2023.05.025. Epub 2023 May 20. PMID 37211143